CLINICAL TRIAL: NCT05124574
Title: Prospective Evaluation of Transplacental Transmission of SARS-COV-2 (COVID-19) in a Cohort of 10 Mother/Child Dyads
Brief Title: Transplacental Transmission of COVID-19
Status: Terminated | Type: Observational
Why Stopped: No cases of COVID recorded in maternity wards since April 2022
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1362021
Record Dates: First submitted 2021-11-16; First posted 2021-11-18 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: SARS-COV-2 Infection
Keywords: immune response; SARS-COV-2; ACE2 receptors; MPRSS2; cathepsin L
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PCR nasopharyngeal, blood (serology SARS-COV-2 and RT-qPCR), placental tissues (see details)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- mothers infected with SARS-COV-2 at the time of delivery.: Maternal-fetal transmission of SARS-COV-2 is likely and may require co-expression of the virus receptor (ACE2) and at least one activator of virus internalization (TMPRSS2 and/or cathepsin) in a cell to make it susceptible to SARS-COV-2 infection.
  To confirm these hypotheses, it is necessary to explore these mechanisms of fetal transmission in a larger number of mothers infected with SARS -CoV-2 at the time of delivery.
  Informed information will be given in the delivery room, initially orally by the midwives, to any mother presenting with an SARS-COV-2 infection (symptomatic or not) (whatever the variant involved). An information leaflet will also be given to the patient and consent will be systematically obtained.
  Interventions: Other: Samples concern SARS-COV-2 + pregnant women at the time of childbirth; Other: Samples concern newborns of SARS-COV-2 + mothers at birth

INTERVENTIONS:
Other: Samples concern SARS-COV-2 + pregnant women at the time of childbirth — * nasopharyngeal PCR in the mother (performed systematically in this epidemic context),
  * Blood samples: 1 EthyleneDiamineTetraacetic Acid (EDTA) tube (immunohistochemistry), 1 yellow tube (COVID + RT-qPCR serology).
  * Sampling of amniotic fluid in case of cesarean section
  * Sampling of the placenta for histological and virological study.
Other: Samples concern newborns of SARS-COV-2 + mothers at birth — * In the birth room:
    * Collection of gastric fluid (PCR SARS-COV-2),
    * Cord blood: 1 EDTA tube (immunohistochemistry), 1 yellow tube (SARS-COV-2 + RT-qPCR serology).
  * In the newborn at D3 of life:
    - 1 yellow tube (SARS-COV-2 + RT-qPCR serology) at the same time as the DNN.
  * In symptomatic newborns:
    * 1 yellow tube (SARS-COV-2 + RT-qPCR serology).
    * nasopharyngeal PCR,

SUMMARY:
SARS-CoV-2, the agent responsible for pandemic COVID-19 infection, is transmitted mainly by respiratory droplets. Regarding maternal-fetal transmission, even if the mode of transmission from mother to fetus is not clear, some cases of perinatal transmission have been described, but without certainty on the routes of placental contamination, trans-cervical or by environmental exposure. .

The case described by J. Vivanti of a newborn with neonatal neurological involvement and whose mother had been infected during the last trimester of pregnancy reports possible transplacental transmission in a context of positive and elevated viremia in the mother and positive viremia in the newborn.

DETAILED DESCRIPTION:
In 2021, it becomes essential to clarify if and how SARS-COV-2 reaches the fetus, in order to prevent neonatal infection, optimize pregnancy management and better understand the pathogenesis of COVID-19.

SARS-COV-2, ACE2 and TMPRSS2 co-receptors are highly expressed in placental tissues and may be actively involved in transplacental transmission of the virus. From a case of materno-fetal transmission described by our team (publication in progress), we observed placental expression of the Spike SARS-COV-2 protein, but also of the ACE2 receptors, TMPRSS2 and cathepsin L. Cytotrophoblast and syncytiotrophoblast cell stains were positive within the placental villi. Maternal leukocytes were also labeled for these proteins.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Signed informed consent
* Pregnant woman with proven SARS-COV-2 infection during full-term delivery

Exclusion Criteria:

* Patient vaccinated within 15 days prior to inclusion

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant woman with proven SARS-COV-2 infection during full-term delivery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Spike SARS-COV-2 protein in placental tissues | Baseline : childbirth
  number of cells expressing the Spike SARS-COV-2 protein

SECONDARY OUTCOMES:
ACE2 receptors in placental tissues | Baseline : childbirth
  number of cells expressing the ACE2 receptors
TMPRSS2 in placental tissues | Baseline : childbirth
  number of cells expressing the TMPRSS2
cathepsin L in placental tissues | Baseline : childbirth
  number of cells expressing the cathepsin L

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No